CLINICAL TRIAL: NCT06815822
Title: Prevention of Postoperative Hernias in Emergency Surgery
Acronym: PROPHECY
Status: Recruiting | Type: Observational
Sponsor: Jan Kochanowski University (Other)
Responsible Party: Principal Investigator, Bartosz Molasy, MD, PhD, Jan Kochanowski University
Other Study IDs: CMUJK 5/2025
Record Dates: First submitted 2025-02-03; First posted 2025-02-07 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-05

CONDITIONS: Incarcerated Hernia; Appendicitis Acute; Cholecystitis, Acute; Ileus; Perforated Gastro-duodenal Ulcers; Perforated Bowel
Keywords: postoperative hernia; trocar site hernia; parastomal hernia; incisional hernia; outcomes; emergency surgery
MeSH Terms: conditions — Appendicitis; Cholecystitis, Acute; Ileus; Intestinal Perforation; Incisional Hernia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Laparotomy: Patients undergoing surgery for acute appendicitis/acute cholecystitis/incarcerated hernia/gastrointestinal perforation or obstruction via laparotomy.
- Laparoscopic/robotic: Patients undergoing surgery for acute appendicitis/acute cholecystitis/incarcerated hernia/gastrointestinal perforation or obstruction via laparoscopy or robotic surgery.

SUMMARY:
The aim of this observational study is to understand the risk factors and incidence of postoperative hernias among patients undergoing emergency surgery. The main question it aims to answer is:

What is the incidence of postoperative hernias in this group of patients?

A brief telephone interview will be conducted with participants who will be included in this study one year after the surgery. If the presence of a postoperative hernia is suspected, the patient will be invited to a follow-up visit to the surgical clinic, where the diagnosis will be confirmed by imaging tests.

DETAILED DESCRIPTION:
Introduction Emergency and urgent surgical procedures carry a high risk of complications. One of the long-term complications is postoperative hernia. Despite numerous studies analysing methods to reduce the incidence of this complication, it remains a significant surgical problem. Studies covering both elective and emergency procedures report that postoperative hernias occur in 2% to 40% of operated patients. The discrepancies in reported incidence rates may result from the asymptomatic nature of some hernias. An example is port-site hernias, for which the exact incidence is not fully determined. Another significant surgical issue is parastomal hernias, occurring in up to 50% of patients. Differences in the incidence of postoperative hernias also arise from the method and duration of patient follow-up. Due to these factors and the specificity of emergency procedures, the frequency of postoperative hernias is often underestimated in this patient group.

Considering the clinical consequences of postoperative hernias, preventing their occurrence is crucial. According to the literature, patients with diabetes, chronic lung disease, smoking habits, obesity, immunodeficiency, or a history of previous abdominal surgeries are at high risk of developing postoperative hernias. The European Hernia Society guidelines highlight the need for further research on methods for preventing postoperative hernias. The surgical approach and technique also influence the incidence of this complication. One of the technical factors is the method of fascial closure. According to the World Society of Emergency Surgery guidelines, the "small bites" technique is suggested for closing midline laparotomies to prevent postoperative hernias and wound complications in emergency surgery; however, the evidence comes from elective procedures. These guidelines emphasise the necessity of conducting prospective studies to confirm the efficacy of this technique in emergency and urgent surgeries. Other aspects of surgical technique, such as suture material, routine use of subcutaneous or intra-abdominal drains, and their impact on postoperative hernia incidence, remain a topic of debate.

The number of large, multicentre studies analysing prevention strategies for this complication is limited, especially concerning postoperative management. According to the available literature, including the European Hernia Society guidelines, the use of abdominal binders and the timing of full activity resumption remain controversial and require further investigation. Another known risk factor for postoperative hernias is surgical site infection, which affects approximately one-third of patients undergoing emergency procedures. A less common but significant surgical complication influencing postoperative hernia development is wound dehiscence, with an estimated incidence of around 4%. Both surgical site infections and wound dehiscence are associated with increased perioperative mortality, making the optimisation of therapeutic strategies to reduce their occurrence essential.

Objective The aim of this study is to determine the incidence of postoperative hernias among patients undergoing emergency surgery and to identify modifiable risk factors for their occurrence. Understanding these factors will help reduce the incidence of this complication and improve treatment outcomes by developing effective preventive strategies for this specific patient group.

Methodology This study will be a nationwide, prospective, cohort, multicentre observational study conducted from 1 June 2025 to 31 December 2026. It will be coordinated by the Department of Surgical Medicine with the Laboratory of Medical Genetics, Medical College, Jan Kochanowski University in Kielce. The study has been approved by the Bioethics Committee of Medical College, Jan Kochanowski University in Kielce (approval number: 5/2025).

The study plan is as follows:

1. Recruitment of study centres - April/May 2025.
2. Patient recruitment - 1 June 2025 - 31 December 2025.
3. Follow-up period - 1 January 2026 - 31 December 2026.
4. Data analysis - January 2027.
5. Publication of study results - February/March 2027.

Inclusion and exclusion criteria:

Inclusion criteria:

* Patient age > 18 years.
* Emergency or urgent surgery.
* Specific surgical indications (acute appendicitis, acute cholecystitis, incarcerated hernia, gastrointestinal perforation, and obstruction).

Exclusion criteria:

* Lack of patient consent.
* Open abdomen technique applied.

The study will analyse data from medical history (comorbidities, previous surgical history) and selected preoperative laboratory tests. The method of fascial closure, use of intra-abdominal and subcutaneous drains, and postoperative management will also be assessed. Additionally, preventive measures for surgical site infections, such as wound irrigation, delayed wound closure, and negative pressure dressings, will be evaluated. The study will also examine preventive measures for postoperative hernias, including abdominal binders/tapes and the timing of full physical activity resumption.

Primary outcomes:

* Incidence of incisional hernia.
* Incidence of port-site hernia after laparoscopy.
* Incidence of parastomal hernia after open/laparoscopic stoma formation.

Secondary outcomes:

* Incidence of surgical site infection.
* Incidence of wound dehiscence.

Follow-up will be conducted via a brief telephone medical interview 12 months after hospital discharge to assess the incidence of postoperative hernias. If a postoperative hernia is suspected, the patient will undergo an outpatient examination, and the presence of a hernia will be confirmed via ultrasound or CT scan. After the follow-up period, each participating centre will submit an anonymised database to the study coordinator, where individual datasets will be consolidated for statistical analysis.

Statistical Analysis

The study will analyse the following data:

* Demographic: age, sex, BMI, comorbidities, ASA score, surgical indication.
* Operative: open vs. minimally invasive technique, type of surgery, fascial closure method, wound irrigation, use of subcutaneous drains, and prophylactic negative pressure dressings.
* Postoperative: prevention strategies for postoperative hernias, time to full physical activity resumption.

The incidence of primary outcomes will be assessed with a 95% confidence interval. The frequency of secondary outcomes (surgical site infection and wound dehiscence) will also be evaluated with a 95% confidence interval. Continuous variables will be presented as median with interquartile range, while categorical variables will be reported as case numbers and percentages. Student's t-test or Wilcoxon test will be used for comparing continuous variables, while the Chi-square test will be applied to categorical data. Univariate and multivariate logistic regression models will be developed to assess hernia risk factors. Relative risk for potential risk factors will also be calculated. A p-value < 0.05 will be considered statistically significant. Statistical analysis will be performed using R software in the RStudio environment.

To estimate the study sample size, a power analysis was conducted. A minimum of 255 cases is required to estimate the postoperative hernia incidence with 5% accuracy and a 95% confidence interval. For port-site hernias, at least 188 cases are needed, while for parastomal hernias, 349 cases are required. The required sample size for surgical site infections is 255 cases, and for wound dehiscence, 93 cases. The total study population will consist approximately 500 patients, which includes an estimated 10% dropout rate.

Authorship Criteria Investigators enrolling at least 40 patients will qualify for "named authorship" (two researchers per centre). Those enrolling 20-40 patients will qualify for "named authorship" (one researcher per centre). Researchers enrolling fewer than 20 patients will be listed under "collaborative authorship".

This study will contribute to the understanding of perioperative management in emergency surgery patients and improve treatment outcomes in this group.

ELIGIBILITY:
Inclusion criteria:

* Patient age > 18 years.
* Emergency or urgent surgery.
* Specific surgical indications (acute appendicitis, acute cholecystitis, incarcerated hernia, gastrointestinal perforation, and obstruction).

Exclusion criteria:

* Lack of patient consent.
* Open abdomen technique applied.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The analyzed population will include adult patients operated on for the most common surgical conditions. Since this will be a multicenter study, the data will include different populations. The analyzed population will be fairly uniform in terms of indications for surgery. The analyzed cases will be diverse in terms of comorbidities, age, and gender.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incisional hernia | From the moment of inclusion until one year from the date of surgery.
  Occurrence of postoperative abdominal hernia in the incision line.
Port-site hernia | From the moment of inclusion until one year from the date of surgery.
  Occurrence of port-site hernia after laparoscopy.
Parastomal hernia | From the moment of inclusion until one year from the date of surgery.
  Occurrence of a parastomal hernia after open/laparoscopic stoma formation

SECONDARY OUTCOMES:
Burst abdomen | From the moment of inclusion in the study until 30 days after surgery.
  Occurrence of burst abdomen after surgery.
Surgical site infection | From the moment of inclusion in the study until 30 days after surgery or 90 days in the case of mesh use (if the primary procedure was repair of an incarcerated hernia or the mesh was placed to prevent postoperative hernia).
  Occurrence of surgical site infection.

CONTACTS AND LOCATIONS:
Overall Officials: Bartosz Molasy, MD, PhD, Principal Investigator — Medical College of the Jan Kochanowski University, Kielce, Poland
Locations (1):
- Department of General Surgery, St Alexander Hospital, Kielce, Poland

IPD SHARING:
Plan to Share IPD: Yes
The IPD will be shared via the Medical College of the Jan Kochanowski University in Kielce website. The shared components will include the study protocol, informed consent form and clinical study report.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: The study protocol and informed consent form will be available before the start of the project. The clinical study report will be available after the end of the project. The IPD will be available for 2 years from the date of the end of the study.
Access Criteria: Access will be open to all interested.

REFERENCES:
- [Background] Kvist M, Jensen TK, Snitkjaer C, Burcharth J. The clinical consequences of burst abdomen after emergency midline laparotomy: a prospective, observational cohort study. Hernia. 2024 Oct;28(5):1861-1870. doi: 10.1007/s10029-024-03104-x. Epub 2024 Jul 20. PMID 39031235
- [Background] Deerenberg EB, Henriksen NA, Antoniou GA, Antoniou SA, Bramer WM, Fischer JP, Fortelny RH, Gok H, Harris HW, Hope W, Horne CM, Jensen TK, Kockerling F, Kretschmer A, Lopez-Cano M, Malcher F, Shao JM, Slieker JC, de Smet GHJ, Stabilini C, Torkington J, Muysoms FE. Updated guideline for closure of abdominal wall incisions from the European and American Hernia Societies. Br J Surg. 2022 Nov 22;109(12):1239-1250. doi: 10.1093/bjs/znac302. PMID 36026550
- [Background] Henriksen NA, Deerenberg EB, Venclauskas L, Fortelny RH, Miserez M, Muysoms FE. Meta-analysis on Materials and Techniques for Laparotomy Closure: The MATCH Review. World J Surg. 2018 Jun;42(6):1666-1678. doi: 10.1007/s00268-017-4393-9. PMID 29322212
- [Background] Goodenough CJ, Ko TC, Kao LS, Nguyen MT, Holihan JL, Alawadi Z, Nguyen DH, Flores JR, Arita NT, Roth JS, Liang MK. Development and validation of a risk stratification score for ventral incisional hernia after abdominal surgery: hernia expectation rates in intra-abdominal surgery (the HERNIA Project). J Am Coll Surg. 2015 Apr;220(4):405-13. doi: 10.1016/j.jamcollsurg.2014.12.027. Epub 2015 Jan 2. PMID 25690673
- [Background] Holihan JL, Alawadi Z, Martindale RG, Roth JS, Wray CJ, Ko TC, Kao LS, Liang MK. Adverse Events after Ventral Hernia Repair: The Vicious Cycle of Complications. J Am Coll Surg. 2015 Aug;221(2):478-85. doi: 10.1016/j.jamcollsurg.2015.04.026. Epub 2015 May 9. PMID 26206646
- [Background] Antoniou SA, Agresta F, Garcia Alamino JM, Berger D, Berrevoet F, Brandsma HT, Bury K, Conze J, Cuccurullo D, Dietz UA, Fortelny RH, Frei-Lanter C, Hansson B, Helgstrand F, Hotouras A, Janes A, Kroese LF, Lambrecht JR, Kyle-Leinhase I, Lopez-Cano M, Maggiori L, Mandala V, Miserez M, Montgomery A, Morales-Conde S, Prudhomme M, Rautio T, Smart N, Smietanski M, Szczepkowski M, Stabilini C, Muysoms FE. European Hernia Society guidelines on prevention and treatment of parastomal hernias. Hernia. 2018 Feb;22(1):183-198. doi: 10.1007/s10029-017-1697-5. Epub 2017 Nov 13. PMID 29134456
- [Background] de Beaux AC, East B. Thoughts on Trocar Site Hernia Prevention. A Narrative Review. J Abdom Wall Surg. 2022 Dec 21;1:11034. doi: 10.3389/jaws.2022.11034. eCollection 2022. PMID 38314166
- [Background] Bosanquet DC, Ansell J, Abdelrahman T, Cornish J, Harries R, Stimpson A, Davies L, Glasbey JC, Frewer KA, Frewer NC, Russell D, Russell I, Torkington J. Systematic Review and Meta-Regression of Factors Affecting Midline Incisional Hernia Rates: Analysis of 14,618 Patients. PLoS One. 2015 Sep 21;10(9):e0138745. doi: 10.1371/journal.pone.0138745. eCollection 2015. PMID 26389785
- [Background] Sanders DL, Pawlak MM, Simons MP, Aufenacker T, Balla A, Berger C, Berrevoet F, de Beaux AC, East B, Henriksen NA, Klugar M, Langaufova A, Miserez M, Morales-Conde S, Montgomery A, Pettersson PK, Reinpold W, Renard Y, Slezakova S, Whitehead-Clarke T, Stabilini C. Midline incisional hernia guidelines: the European Hernia Society. Br J Surg. 2023 Nov 9;110(12):1732-1768. doi: 10.1093/bjs/znad284. No abstract available. PMID 37727928
- [Background] Frassini S, Cobianchi L, Fugazzola P, Biffl WL, Coccolini F, Damaskos D, Moore EE, Kluger Y, Ceresoli M, Coimbra R, Davies J, Kirkpatrick A, Di Carlo I, Hardcastle TC, Isik A, Chiarugi M, Gurusamy K, Maier RV, Segovia Lohse HA, Jeekel H, Boermeester MA, Abu-Zidan F, Inaba K, Weber DG, Augustin G, Bonavina L, Velmahos G, Sartelli M, Di Saverio S, Ten Broek RPG, Granieri S, Dal Mas F, Fare CN, Peverada J, Zanghi S, Vigano J, Tomasoni M, Dominioni T, Cicuttin E, Hecker A, Tebala GD, Galante JM, Wani I, Khokha V, Sugrue M, Scalea TM, Tan E, Malangoni MA, Pararas N, Podda M, De Simone B, Ivatury R, Cui Y, Kashuk J, Peitzman A, Kim F, Pikoulis E, Sganga G, Chiara O, Kelly MD, Marzi I, Picetti E, Agnoletti V, De'Angelis N, Campanelli G, de Moya M, Litvin A, Martinez-Perez A, Sall I, Rizoli S, Tomadze G, Sakakushev B, Stahel PF, Civil I, Shelat V, Costa D, Chichom-Mefire A, Latifi R, Chirica M, Amico F, Pardhan A, Seenarain V, Boyapati N, Hatz B, Ackermann T, Abeyasundara S, Fenton L, Plani F, Sarvepalli R, Rouhbakhshfar O, Caleo P, Ho-Ching Yau V, Clement K, Christou E, Castillo AMG, Gosal PKS, Balasubramaniam S, Hsu J, Banphawatanarak K, Pisano M, Adriana T, Michele A, Cioffi SPB, Spota A, Catena F, Ansaloni L. ECLAPTE: Effective Closure of LAParoTomy in Emergency-2023 World Society of Emergency Surgery guidelines for the closure of laparotomy in emergency settings. World J Emerg Surg. 2023 Jul 26;18(1):42. doi: 10.1186/s13017-023-00511-w. PMID 37496068
- [Derived] Molasy B, Zamkowski M, Mitura K, Smietanski M. Prevention of Postoperative Hernias in Emergency Surgery - PROPHECY Trial. J Abdom Wall Surg. 2025 Jul 9;4:14765. doi: 10.3389/jaws.2025.14765. eCollection 2025. PMID 40703916